CLINICAL TRIAL: NCT06253936
Title: Prevalence of Anatomical Variants of Dural Sinuses by Magnetic Resonance Venography Evaluation in Sohag
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Marina Makram Sabah, Prevalence of anatomical variants of dural sinuses by Magnetic Resonance Venography evaluation in Sohag, Sohag University
Other Study IDs: Soh-Med-24-01-01MS
Record Dates: First submitted 2024-02-04; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Anatomical Variants of Dural Sinuses by Magnetic Resonance Venography

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Magnetic Resonance Venography — Detect the anatomical variants of dural sinuses by Magnetic Resonance Venography

SUMMARY:
MR cerebral venography (MRV) is an MRI examination of the head with either contrast-enhanced or non-contrast sequences to assess patency of the dural venous sinuses and cerebral veins.

ELIGIBILITY:
Inclusion Criteria:

* Sohag by nationality and residence, male or female by sex, having normal cerebral MRV reported and consented to participate in the research work will be included in this research.

Exclusion Criteria:

* Having the diagnosis of cerebral venous sinus thrombosis, and previous head injury are the exclusion criteria of this research, also patients with absolute or relative contraindications for imaging including; claustrophobia, metallic implants, pacemaker and prosthetic heart valves for MRI.

Ages: 7 Days to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Sohag by nationality and residence, male or female by sex, having normal cerebral MRV reported and consented to participate in the research work will be included in this research.
Sampling Method: Probability Sample
Enrollment: 169 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of anatomical variants of dural sinuses by Magnetic Resonance Venography evaluation in Sohag | 1 year
  The primary outcome for the study is to assess the number of anatomical variants of dural sinuses by MRV evaluation among patients attended to Sohag University Hospitals. Standard head coils with small field of view and thin sections will be used for the examination. Routine MRI brain including Axial T1WI, T2WI, FLAIR, Coronal T2WI, and Sagittal T1 WI will be done with complementary Maximum intensity projection (MIP) 3D MR venography. Imaging findings of the veins and sinuses will be recorded using Philips Achieva1.5T MRI device (Philips Achieva, Netherlands) or Siemens Magnetom Altea1.5T MRI device (Siemens Healthineers, Germany). Any anatomic variants in these sinuses or their drainage, if any, will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes